CLINICAL TRIAL: NCT04928599
Title: Financial Distress During Treatment for Pediatric Acute Lymphoblastic Leukemia in the United States
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Other Study IDs: ACCL20N1CD; NCI-2021-03567 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCL20N1CD (Other: Children's Oncology Group); COG-ACCL20N1CD (Other: DCP); ACCL20N1CD (Other: CTEP); UG1CA189955 (NIH)
Record Dates: First submitted 2021-05-04; First posted 2021-06-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Health Services Research (survey, interview, chart review): Parents complete surveys over 15-30 minutes at the beginning of their child's induction chemotherapy, at the beginning of maintenance chemotherapy, and at the end of last chemotherapy. Parents may also participate in one-time individual interview over 30-45 minutes. Additionally, children's medical records are reviewed during the study
  Interventions: Other: Electronic Health Record Review; Other: Interview; Other: Survey Administration

INTERVENTIONS:
Other: Electronic Health Record Review — Review of medical records
Other: Interview — Complete interview
Other: Survey Administration — Complete survey

SUMMARY:
The overall goals of this study are to measure parents' financial distress (worry or anxiety about money) during their child's/adolescent's treatment for acute lymphoblastic leukemia and whether it changes over time, and to learn what factors are associated with changes in financial distress. Information gathered from this study will inform future intervention studies that may mitigate financial distress for parents of children/adolescents being treated for acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the trajectory of financial distress over time, as reported by parents of children and adolescents ages 1 to 14.9 years with acute lymphoblastic leukemia (ALL), from start to completion of ALL therapy.

SECONDARY OBJECTIVE:

I. Identify factors associated with financial distress over time for families of children and adolescents ages 1 to 14.9 years with newly diagnosed ALL.

EXPLORATORY OBJECTIVES:

I. Describe domains of financial toxicity, informed by the conceptual framework guiding this study, specifically treatment-related material hardship during treatment for pediatric ALL, potential financial coping behaviors during treatment for pediatric ALL, and institutional factors.

II. In a sub-cohort of participants, qualitatively explore parental experiences of financial distress and material hardship, and perceptions about financial screening/assessments during their child's/adolescent's treatment for ALL.

OUTLINE: This is an observational study.

Parents complete surveys over 15-30 minutes at the beginning of their child's induction chemotherapy, at the beginning of maintenance chemotherapy, and at the end of last chemotherapy. Parents may also participate in one-time individual interview over 30-45 minutes. Additionally, children's medical records are reviewed during the study.

ELIGIBILITY:
Inclusion Criteria:

* All Children's Oncology Group (COG) NCI Community Oncology Research Program (National Cancer Institute [N]CORP) institutions are eligible for participation in this study upon first parent enrollment
* Parents of an index child who meets the following characteristics are eligible for this study:

  * Index child must be newly diagnosed with de novo ALL
  * Index child must be between the ages of 1 and 14.9 years at the time of the parent's enrollment
  * At the parent's entry to the study, the index child must be receiving induction chemotherapy for newly diagnosed ALL at the enrolling institution. The index child may be enrolled in therapeutic clinical ALL trials or receiving ALL therapy per standard of care
* Parents age 18 years and above are eligible for this study
* Parent must speak English or Spanish in order to participate in the consent process and provide consent. The parent's language skills must be sufficient to understand the study requirements and complete the survey and interview questions
* At the parent's entry to the study, the index child must be receiving induction chemotherapy for newly diagnosed ALL at the enrolling institution. The index child may be enrolled in therapeutic clinical ALL trials or receiving ALL therapy per standard of care
* REGULATORY REQUIREMENTS: All parents must sign a written informed consent for their participation in the study
* REGULATORY REQUIREMENTS: All institutional and NCI requirements for human studies must be met

Exclusion Criteria:

* Parents of index children with any of the following clinical characteristics will be excluded from the study:

  * KMT2A-R (formerly MLL-R) not receiving ALL therapy
  * Mixed-phenotype acute leukemia (MPAL) not receiving ALL therapy
  * Burkitt's leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents of children who are receiving induction chemotherapy for newly diagnosed ALL
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in financial distress | From start through completion of acute lymphoblastic leukemia therapy, an average of 2.5 years
  Financial distress will be measured serially using the Personal Finance Wellbeing (PFW) scale (previously InCharge Financial Distress/Financial Well-Being scale). Scores on the PFW scale will be computed by adding numerical responses for each of the 8 questions, then dividing the total by 8. These scores can range from 1 to 10, with 1 indicating overwhelming financial distress and 10 indicating no financial distress.

SECONDARY OUTCOMES:
Factors associated with financial distress | From start of through completion of acute lymphoblastic leukemia therapy, an average of 2.5 years
  Candidate factors include socio-demographic variables, clinical variables, institutional variables, financial variables (e.g., Household Material Hardship [HMH] scores, change in household income), and financial coping behaviors.

OTHER OUTCOMES:
Domains of financial toxicity | From start through completion of acute lymphoblastic leukemia therapy, an average of 2.5 years
  Descriptive statistics will be used to report domains of financial distress, informed by the conceptual framework guiding this study.
Parental experiences of financial distress and material hardship, and perceptions about financial screening/assessments during their child's/adolescent's treatment | From start through completion of acute lymphoblastic leukemia therapy, an average of 2.5 years
  Each audio-recorded interview, and the associated field notes and summary, will be transcribed verbatim. These data will be coded using a directed content analysis approach.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa P Beauchemin, Principal Investigator — Children's Oncology Group
Locations (40):
- United States (39):
  - Kaiser Permanente-Oakland, Oakland, California
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Blank Children's Hospital, Des Moines, Iowa
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Morristown Medical Center, Morristown, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Geisinger Medical Center, Danville, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
- University Pediatric Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Beauchemin M, Santacroce SJ, Bona K, Dang H, Alexander S, Allen K, De Los Santos C, Fisher B, Muneton-Castano Y, Ponce O, Vargas S, Sugalski A, Sung L, Parsons S. Rationale and design of Children's Oncology Group (COG) study ACCL20N1CD: financial distress during treatment of acute lymphoblastic leukemia in the United States. BMC Health Serv Res. 2022 Jun 28;22(1):832. doi: 10.1186/s12913-022-08201-0. PMID 35764995